CLINICAL TRIAL: NCT07215741
Title: A Retrospective, Multi-center Real-world Study of StimLabs Human Placental Membrane Tissue Used for Treatment in Hard-to-Heal Wounds
Brief Title: Retrospective, Multi-center Real-world Study of StimLabs Human Placental Membrane Tissue to Treat Hard-to-Heal Wounds
Status: Active, not recruiting | Type: Observational
Sponsor: StimLabs (Industry)
Responsible Party: Sponsor
Other Study IDs: REL2501.000-M (07/25)
Record Dates: First submitted 2025-09-25; First posted 2025-10-10 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-09

CONDITIONS: Chronic Wounds; Diabetic Ulcers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Retrospective Relese: Retrospective case review to include all subjects that received Relese between May 2023 to April 2025.

SUMMARY:
This is a retrospective, multi-center observational study to assess real-world outcomes of StimLabs human placental membrane tissue used in the treatment of hard-to-heal wounds, including chronic ulcers, diabetic foot ulcers (DFUs), and venous leg ulcers (VLUs). The collection of retrospective real-world data provides a broad range of experiences related to patient healthcare and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive diabetic subjects that received a Relese product application during treatment between May 2023 and April 2025.

Exclusion Criteria:

* Subjects not receiving an initial Relese application during treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive subjects receiving Relese in a real-world setting
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The proportion of target ulcers achieving complete wound closure during the observational period | 1-12 weeks
  Determine the percent (%) of target ulcers achieving complete wound closure at 12 weeks.

SECONDARY OUTCOMES:
Percent area reduction | 1-12 weeks
  Percent Area Reduction (PAR) will be calculated from Treatment Visit 1 to Treatment Visit 12.
Time to closure for the target ulcer | 1-12 weeks
  Time to closure (days) will be determined from the first product application to the date when the wound is first documented as fully closed.
Adverse events | 1-12 weeks
  Incidence of adverse events will be evaluated weekly.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Cypress Wound Care, Oklahoma City, Oklahoma
  - Premier Foot & Ankle, Denison, Texas
  - Premier Foot & Ankle, Frisco, Texas